CLINICAL TRIAL: NCT03838783
Title: Flexible Insulin Therapy Untethered Insulin Regimen Using Insulin Degludec and Continuous Subcutaneous Insulin Infusion in Avidly Exercising Patients With Type 1 Diabetes: FIT Untethered
Brief Title: Flexible Insulin Therapy Untethered Insulin Regimen in Avidly Exercising Patients With Type 1 Diabetes: FIT Untethered
Acronym: FIT Untethered
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LMC Diabetes & Endocrinology Ltd. (Other)
Responsible Party: Principal Investigator, Ronnie Aronson, MD, Chief Medical Officer, LMC Diabetes & Endocrinology Ltd.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FIT Untethered
Record Dates: First submitted 2018-07-26; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Exercise; Insulin Degludec; Continuous glucose monitoring (CGM); Continuous Subcutaneous Insulin Infusion (CSII)
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity | interventions — insulin degludec

STUDY DESIGN:
Intervention Model Description: Randomization for the sequence of Interventions (A and B) will be done by an interactive system that will randomly assign patients to an intervention sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual CSII (No Intervention): Continue to use the established CSII insulin therapy
- Untethered CSII (Experimental): Basal dosing - total CSII basal dose will be delivered by 50% through continuing CSII therapy used prior to study enrollment and 50% through the addition of once daily insulin degludec injected in the morning; Bolus dosing - continue the established bolus insulin dose
  Interventions: Drug: Insulin Degludec

INTERVENTIONS:
Drug: Insulin Degludec — 50% of the patient's daily basal insulin dose delivered through once daily insulin degludec injected in the morning; 50% of the basal insulin to be delivered through previously established CSII
  Other Names: Tresiba
  Arms: Untethered CSII

SUMMARY:
The overall objective of this study is to evaluate glycemic control and patient-reported outcomes in patients with Type 1 diabetes (T1D) who use insulin degludec and continuous subcutaneous insulin infusion in a combination untethered regimen during moderate or high-intensity exercise.

DETAILED DESCRIPTION:
FIT untethered is an open-label, randomized, repeated measures cross-over design study, testing glycemic control in "untethered" continuous subcutaneous insulin infusion (CSII) therapy compared to usual CSII therapy, in physically active patients with T1D (N=30). During 2-week screening visits, participants are randomized into either the usual CSII arm or the untethered CSII arm. Patients in the usual group continue with their established CSII therapy. Patients in the untethered group are to administer 50% of their basal dose through an insulin degludec injection every morning, with the other 50% achieved through their established CSII therapy. Bolus insulin remains at the established dose in both groups. After randomization, patients begin Phase I and transition into a 2-week insulin optimization period. Then, participants will complete 2 in-clinic, supervised exercise visits (1 moderate and 1 high intensity exercises) in the following week. After, participants must complete 2 unsupervised at-home exercises per week for 3 weeks (cumulative total of 2 moderate and 4 high intensity exercises). After the home exercise period, participants cross-over to the other study arm and begin Phase II. Phase II is similar to Phase I: 2 weeks of insulin dose optimization, 1 week of supervised clinic exercise, and 3 weeks of unsupervised home exercise. For both in-clinic and home-based exercise, the participant's insulin pump will be disconnected and suspended 60 minutes prior to beginning the workout, and will be reconnected immediately following each workout. A continuous glucose monitoring (CGM) device will be worn by each participant for the entire duration of the study. The co-primary outcomes of the study include time in range (4.0 - 10.0 mmol/L) in the 6 hours after the start of moderate- and high-intensity exercise. The key secondary outcomes include the glucose variability during the 24 hour period after the start of both moderate and high intensity exercise, and patient reported outcomes before and after exercise.

ELIGIBILITY:
Inclusion Criteria:

* Adults with clinical diagnosis of T1D
* Age 18-55 years, inclusive
* Diagnosis of T1D ≥ 6 months
* A1c ≤ 8.5% at screening visit
* Using stable CSII therapy for ≥ 6 months
* Exercise regularly (≥ 3 times per week of moderate or vigorous exercise)
* VO2peak ≥ 30 ml/kg/min for females and ≥ 32 ml/kg/min for males
* Willing to adhere to the protocol requirements for the duration of the study
* Written informed consent
* Fasting C-peptide value of < 0.7 ng/mL (0.23 nmol/L) at screening visit

Exclusion Criteria:

* Pregnant or lactating
* Already using a split regimen of combination CSII and basal insulin injection
* Active diabetic retinopathy (proliferated diabetic retinopathy, or vitreous hemorrhage in past 6 months) that could potentially be worsened by the exercise protocol
* Any evidence of unstable cardiovascular disease, disorders or abnormalities as per physician's discretion
* Currently following a very low calorie or other weight-loss diet which may impact glucose control and mask the primary and secondary outcome measures
* More than one episode of severe hypoglycemia with seizure, coma or requiring assistance of another person during the past 6 months
* Known hypoglycemia unawareness
* Use of acetaminophen (Tylenol) during the study period
* Medications other than insulin that might impact outcome measures:

  * Beta blockers
  * Any agents that affect hepatic glucose production, including all beta adrenergic agonists or antagonists, all xanthine derivatives
  * Pramlintide
  * Any non-insulin diabetes therapy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Time in range within 6 hours | 6 hours
  Percentage of time with CGM glucose between 4.0 - 10.0 mmol/L within 6 hours after the start of high-intensity or moderate-intensity, in-clinic exercise

SECONDARY OUTCOMES:
Change in glucose within 60 mins after high-intensity exercise starts | 60 mins
  Plasma glucose at 30 mins after after the end of a 30-min high-intensity, in-clinic exercise minus plasma glucose at baseline (right before exercise)
Change in glucose within 120 mins after moderate-intensity exercise starts | 120 mins
  Plasma glucose at 30 mins after the end of a 90-min moderate-intensity, in-clinic exercise minus plasma glucose at baseline (right before exercise)
Time spent in hypoglycemia 24 hours after exercise | 24 hours
  Percentage of time with CGM glucose <4.0 mmol/L within 24 hour after the start of high intensity exercise or moderate intensity in-clinic exercise
Time in range 24 hours after exercise | 24 hours
  Percentage of time with CGM glucose between 4.0 - 10.0 mmol/L within 24 hour after the start of high intensity exercise or moderate intensity in-clinic exercise
Time spent in hyperglycemia 24 hours after exercise | 24 hours
  Percentage of time with CGM glucose > 10.0 mmol/L within 24 hour after the start of high intensity exercise or moderate intensity in-clinic exercise
Time in range in the last 4 weeks of each study phase | 4 weeks
  Percentage of time with CGM glucose between 4.0 - 10.0 mmol/L in the last 4 weeks of each study phase
Frequency of hypoglycemia 24 hours after exercise | 24 hours
  Number of hypoglycemic episodes, which are defined as CGM glucose <4.0 mmol/L lasting ≥15 minutes within 24 hours following high intensity exercise or moderate intensity in-clinic exercise
Frequency of hypoglycemia in the last 4 weeks of each study phase | 4 weeks
  Number of hypoglycemic episodes, which are defined as CGM glucose <4.0 mmol/L lasting ≥15 minutes in the last 4 weeks of each study phase
Change in Diabetes Medication Satisfaction (DiabMedSat) Score | 11 weeks
  Diabetes Medication Satisfaction questionnaire is to measure the level of patients' satisfaction with their diabetes medication(s) in the past 2 weeks. The score range will be 0 to 100. The higher the score, the less the satisfaction.
  The change of scores is the score difference between Visit 24 and Visit 2
Change in Hypoglycemia Fear Score | 11 weeks
  Hypoglycemia Fear will be measured by the Hypoglycemia Fear Survey which assesses the subject's behaviors to avoid hypoglycemia and to measure the subjects' worries about hypoglycemia and its consequences in the past 3 months. The range of the score will be 0 to 132. The higher the score, the greater the fear.
  The changes of scores are the score difference between Visit 24 and Visit 2
Change in TRIM-D Score | 11 weeks
  Treatment Related Impact Measure - Diabetes Device (TRIM-D Device) questionnaire will be used to generate TRIM-D-Score. It measures the level of the subject's satisfaction with the device used to take the diabetes medication. The range of this score will be 3-15. The higher the score, The greater satisfaction.
  The changes of scores are the score difference between Visit 24 and Visit 2

CONTACTS AND LOCATIONS:
Locations (1):
- LMC Diabetes & Endocrinology Ltd., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doyle EA, Weinzimer SA, Steffen AT, Ahern JA, Vincent M, Tamborlane WV. A randomized, prospective trial comparing the efficacy of continuous subcutaneous insulin infusion with multiple daily injections using insulin glargine. Diabetes Care. 2004 Jul;27(7):1554-8. doi: 10.2337/diacare.27.7.1554. PMID 15220227
- [Background] Binek A, Rembierz-Knoll A, Polanska J, Jarosz-Chobot P. Reasons for the discontinuation of therapy of personal insulin pump in children with type 1 diabetes. Pediatr Endocrinol Diabetes Metab. 2016 Feb 18;21(2):65-9. doi: 10.18544/PEDM-21.02.0026. PMID 26901138
- [Background] Wong JC, Boyle C, DiMeglio LA, Mastrandrea LD, Abel KL, Cengiz E, Cemeroglu PA, Aleppo G, Largay JF, Foster NC, Beck RW, Adi S; T1D Exchange Clinic Network. Evaluation of Pump Discontinuation and Associated Factors in the T1D Exchange Clinic Registry. J Diabetes Sci Technol. 2017 Mar;11(2):224-232. doi: 10.1177/1932296816663963. Epub 2016 Sep 25. PMID 27595711
- [Background] Benbenek-Klupa T, Matejko B, Klupa T. Metabolic control in type 1 diabetes patients practicing combat sports: at least two-year follow-up study. Springerplus. 2015 Mar 17;4:133. doi: 10.1186/s40064-015-0919-5. eCollection 2015. PMID 25825689
- [Background] Delvecchio M, Zecchino C, Salzano G, Faienza MF, Cavallo L, De Luca F, Lombardo F. Effects of moderate-severe exercise on blood glucose in Type 1 diabetic adolescents treated with insulin pump or glargine insulin. J Endocrinol Invest. 2009 Jun;32(6):519-24. doi: 10.1007/BF03346499. PMID 19474521
- [Background] Yardley JE, Zaharieva DP, Jarvis C, Riddell MC. The "ups" and "downs" of a bike race in people with type 1 diabetes: dramatic differences in strategies and blood glucose responses in the Paris-to-Ancaster Spring Classic. Can J Diabetes. 2015 Apr;39(2):105-10. doi: 10.1016/j.jcjd.2014.09.003. Epub 2014 Dec 6. PMID 25492557
- [Background] Riddell MC, Gallen IW, Smart CE, Taplin CE, Adolfsson P, Lumb AN, Kowalski A, Rabasa-Lhoret R, McCrimmon RJ, Hume C, Annan F, Fournier PA, Graham C, Bode B, Galassetti P, Jones TW, Millan IS, Heise T, Peters AL, Petz A, Laffel LM. Exercise management in type 1 diabetes: a consensus statement. Lancet Diabetes Endocrinol. 2017 May;5(5):377-390. doi: 10.1016/S2213-8587(17)30014-1. Epub 2017 Jan 24. PMID 28126459
- [Derived] Aronson R, Li A, Brown RE, McGaugh S, Riddell MC. Flexible insulin therapy with a hybrid regimen of insulin degludec and continuous subcutaneous insulin infusion with pump suspension before exercise in physically active adults with type 1 diabetes (FIT Untethered): a single-centre, open-label, proof-of-concept, randomised crossover trial. Lancet Diabetes Endocrinol. 2020 Jun;8(6):511-523. doi: 10.1016/S2213-8587(20)30114-5. PMID 32445738